CLINICAL TRIAL: NCT06769399
Title: Investigation of the Relationship Between Pelvic Floor Dysfunctions and Sexual Dysfunction in Female Patients with Systemic Sclerosis: a Cross-Sectional Study
Brief Title: Relationship Between Pelvic Floor Dysfunctions and Sexual Dysfunction in Female Patients with Systemic Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tulay Ulku SEVIM, Lecturer, Istanbul University - Cerrahpasa
Other Study IDs: 142198O
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Systemic Sclerosis (SSc); Sexual Dysfunctions; Pelvic Floor Disorder
Keywords: systemic sclerosis; female sexual dysfunction; pelvic floor disorders
MeSH Terms: conditions — Scleroderma, Systemic; Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- study group: Female patients with systemic sclerosis
- Control group: healthy women

SUMMARY:
Relationship Between Pelvic Floor Dysfunctions and Sexual Dysfunction in Female Patients with Systemic Sclerosis

DETAILED DESCRIPTION:
Female patients with systemic sclerosis have a high incidence of pelvic floor dysfunction and sexual dysfunction.The association of sexual dysfunction in systemic sclerosis with many disease-related factors has been confirmed. There are numerous studies in the literature investigating the prevalence and risk factors of sexual dysfunction in women with SSc, the number of studies examining the prevalence and effects of pelvic floor dysfunction in SSc is limited. Moreover, no studies were identified in the literature that specifically investigate the relationship between pelvic floor dysfunction and sexual dysfunction.The aim of this study is to evaluate pelvic floor dysfunction and sexual dysfunction in women with SSc, examine the relationship between these dysfunctions, and compare the findings with data from a healthy control group.

ELIGIBILITY:
Inclusion Criteria:

* female gender
* being between 18-64 years old
* having a diagnosis of systemic sclerosis (SSc)
* being sexually active, and not having entered menopause

The control group will consist of healthy women aged 18-64 years who are sexually active, have not entered menopause, have no history of urological or gynecological surgeries other than cesarean section, and have no rheumatologic or severe chronic diseases.

Exclusion Criteria:

* the presence of current or past rheumatologic diseases other than SSc
* the presence of current urogynecological diseases
* a history of urological or gynecological surgeries other than cesarean section.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Study Population: 70 women with systemic sclerosis and 70 healthy women
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
pelvic floor dysfunction | 1 day
  Pelvic Floor Distress Inventory-20 (PFDI-20) will be used.The PFDI-20 is comprised of 3 scales, which include the Urinary Distress Inventory-6 (UDI-6), Pelvic Organ Prolapse Distress Inventory-6 (POPDI-6), and the Colorectal-Anal Distress Inventory-8 (CRADI-8).Since it is comprised of the UDI-6, POPDI-6, and the CRADI-8, the PFDI-20 includes 20 questions. Each question begins with a "yes" or "no" response. If "yes," the patient must indicate how much bowl, bladder, or pelvic symptoms have been bothering them in the past 3 months on a 4-point scale that ranges from "not at all" (0) to "quite a bit" (4). The scale scores are found individually by calculating the mean value of their corresponding questions and then multiplying by 25 to obtain a value that ranges from 0 to 100. The sum of the 3 scales are added together to get the PFDI-20 summary score, which ranges from 0 to 300.
sexual dysfunction | 1 day
  Female Sexual Function Index (FSFI) will be used.The FSFI is a 19-item patient-reported outcome measure, consisting of 6 separate domains of female sexual function, namely desire (items 1-2), arousal (3-6), lubrication (7-10), orgasm (11-13), satisfaction (14-16), and pain (17-19).Total scores range from 2-30 with lower scores corresponding to worse sexual functioning.
Pelvic Floor Dysfunction | 1 day
  Pelvic Floor Impact Questionnaire-7(PFIQ-7). It is a health-related quality of life questionnaire for women with pelvic floor conditions to fill out. It includes scales from the Urinary Impact Questionnaire (UIQ-7), Pelvic Organ Prolapse Impact Questionnaire (POPIQ-7), and the Colorectal-Anal Impact Questionnaire-7 (CRAIQ-7), which are short-forms of their the longer versions.The PFIQ-7 consists of 7 questions that need to be answered 3 times each considering symptoms related to the bladder or urine, vagina or pelvis, and bowel or rectum and their effect on function, social health, and mental health in the past 3 months.The scale scores are then added together to get the total PFIQ-7 score, which ranges from 0-300. A lower score means there is a lesser effect on quality of life.

SECONDARY OUTCOMES:
Functional Capacity | 1 day
  Scleroderma Health Assessment Questionnaire will be used.
disease activity | 1 day
  Modified Rodnan Skin Score will be used.

IPD SHARING:
Plan to Share IPD: No